CLINICAL TRIAL: NCT00701636
Title: Pharmacokinetics of Daptomycin During Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry); Hartford Hospital (Other); Western University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12903-01; IIS 0003-07-2007 (Other: Cubist Pharmaceuticals)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Late Effects of Surgery; Staphylococcus Aureus; Surgical Site Infection
Keywords: Daptomycin; Antibiotic Prophylaxis; Pharmacokinetics; Surgical Wound Infection; Staphylococcus aureus; Cardiopulmonary Bypass Surgery
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cases (Experimental): The first 15 subjects enrolled will receive the intervention drug daptomycin as surgical antibiotic prophylaxis.
  Interventions: Drug: daptomycin
- Controls (No Intervention): 15 subjects will be enrolled in the standard of care antibiotic group to serve as the controls. Controls will receive no experimental medications or treatments. The purpose of enrolling control patients was to serve as a reference group for intervention patients. Specifically cases and controls will be compared for changes in commonly collected hematologic parameters, creatinine, and CPK. Additionally, parameters collected during anesthesia will be compared. Controls will be matched to the intervention group by age (+/- 10 years), gender, and ethnicity.

INTERVENTIONS:
Drug: daptomycin — Subjects enrolled in the intervention group will receive a single intravenous administration of daptomycin 8 mg/kg 30-60 minutes prior to surgery (incision). The 500 mg vial will be reconstituted with 10 mL of 0.9% normal saline (NS) and further diluted in 50 mL of 0.9% NS to be given over a 30 minute infusion.
  Other Names: Cubicin
  Arms: Cases

SUMMARY:
This investigation is a prospective, open-label pharmacokinetic study of daptomycin prophylaxis in patients undergoing coronary artery bypass graft surgery without valvular replacement.

DETAILED DESCRIPTION:
Cardiothoracic surgery is a commonly performed procedure in the United States. Many sites previously used cefazolin, an antibiotic, as standard prophylaxis to prevent surgical site infections. However, given most bacteria causing surgical site infections are now resistant to cefazolin, most center are using vancomycin, an alternative antibiotic, as surgical antibiotic prophylaxis. However, some patients cannot take vancomycin, and there are no well studied alternatives to vancomycin for surgical prophylaxis. Therefore, we are studying daptomycin, a newer United States Food and Drug Administration (FDA)-approved antibiotic, as prophylaxis against surgical site infections among patients undergoing cardiothoracic bypass (CPB) with coronary artery bypass graft surgery (CABG). Our study will not be powered to see if daptomycin is as effective as vancomycin at preventing surgical site infections. Instead, the purpose of this study is to validate that adequate levels of antibiotics are present in patients' blood during cardiothoracic bypass surgery.

Study subjects in the intervention group will be followed from the time of enrollment in the study until their discharge from the hospital, or up to 7 days following administration of daptomycin, whichever comes first.

The first 15 subjects enrolled will receive the intervention drug daptomycin as surgical antibiotic prophylaxis and the following 15 subjects will be enrolled as matched controls and will receive the standard of care surgical prophylaxis per the patient's treating physicians. The controls will undergo monitoring for the same safety outcomes that the patients who received daptomycin will undergo.

Subjects enrolled in the intervention group will receive a single intravenous administration of daptomycin 8 milligram (mg)/kilogram (kg) 30-60 minutes prior to surgery (incision). Blood samples will be drawn by the Research Coordinator. A total of 85 (milliliters) mL of blood will be collected during the study. A total of 14 blood samples will be collected: 4 samples at the Pre-CPB phase, 4 samples during the CPB procedure, and 6 samples Post-CPB. Total plasma daptomycin concentrations will be determined utilizing standard high-performance liquid chromatography techniques. Plasma concentrations will be compared to the minimum inhibitory concentrations (MIC90) of the common pathogens involved in surgical site infections, specifically Staphylococcus aureus and coagulase negative Staphylococcus.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients, awaiting scheduled elective coronary artery bypass graft (CABG) surgery without valve replacement surgery
* Age > 18 years and < 75 years
* BMI between 18.5 and 35.0 kg/meters-squared
* Crcl > 50 ml/minute calculated based on Cockcroft Gault equation
* No known active or suspected infection(s)
* Ability to complete the informed consent process
* Negative pregnancy test (for women of childbearing age)

Exclusion Criteria:

* History of allergic reaction to daptomycin or components of daptomycin
* Receipt of daptomycin within 7 days prior to the surgery
* Elevated CPK levels (defined as > 3 times the upper limits of known normal)
* History of myopathy or complaints consistent with myopathy
* Current or planned use of mycophenolate mofetil, mycophenolic acid, or tobramycin during the subjects' current hospitalization (all of which are known to interact with daptomycin)
* Inability to complete the informed consent process because of problems with mental capacity
* Pregnancy and/or breast feeding

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren G Miller, M.D., M.P.H., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared upon written request to the principal investigator.

REFERENCES:
- [Result] Nguyen MH, Eells SJ, Tan J, Sheth CT, Omari B, Flores M, Wang J, Miller LG. Prospective, open-label investigation of the pharmacokinetics of daptomycin during cardiopulmonary bypass surgery. Antimicrob Agents Chemother. 2011 Jun;55(6):2499-505. doi: 10.1128/AAC.01404-10. Epub 2011 Mar 28. PMID 21444695
- See also: Free full text article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3101392/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2008 to August 2010, we recruited subjects undergoing CABG surgery at Harbor-UCLA Medical Center, a 400-bed tertiary-care county hospital.
Period: Overall Study
Arm/Group | Cases | Controls
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Our protocol says we will enroll 32 subjects, with the assumption that 2 may not finish the study, have protocol violations, or have data that is corrupt and unusable. Our target was 30 analyzable subjects. Since we had no subjects withdraw from the trial, and no protocol violations or data problems, we halted enrollment at 30 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8.0) | 57 (8.7) | 56 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Daptomycin Concentrations at 12, 18, 24, and 48 h
Description: Mean daptomycin concentrations (mcg/ml) at 12, 18, 24, and 48 h
Time Frame: Hospital discharge or 7 days, whichever comes first
Population: Based on sample sizes from previously published studies on antibiotic pk for CABG surgery.
Measure: Mean (Standard Deviation); unit: mcg/ml
Groups:
- Cases: The first 15 subjects enrolled will receive the intervention drug daptomycin as surgical antibiotic prophylaxis for CABG.
Arm/Group | Cases
Number analyzed (Participants) | 15
mcg/ml
  mean daptomycin concentration at 12 hours | 22.7 (9.7)
  mean daptomycin concentration at 18 hours | 16.2 (8.2)
  mean daptomycin concentration at 24 hours | 12.0 (4.7)
  mean daptomycin concentration at 48 hours | 3.5 (2.3)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cases | Controls
Serious Adverse Events (participants affected / at risk) | 0/15 | 3/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cases (N=15) | Controls (N=15)
Surgical site infection (Surgical and medical procedures) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No